CLINICAL TRIAL: NCT00380835
Title: A Phase 2 Trial of Amrubicin With or Without Herceptin in the Treatment of Metastatic Breast Cancer
Brief Title: Study of Amrubicin With or Without Herceptin in Patients With Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Never Initiated
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNF3140-MBC-001
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; amrubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — amrubicin

INTERVENTIONS:
Drug: Amrubicin

SUMMARY:
The purpose of the study is to evaluate the incidence of cardiac toxicity of amrubicin when administered to patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of breast cancer.
* Metastatic or recurrent disease, either HER2+ (FISH+ or 3+ IHC) or HER2-.
* Maximal dose of prior adjuvant anthracycline: 300 mg/meters squared doxorubicin or equivalent. Relapse greater than one year after trastuzumab adjuvantly; two years following adjuvant anthracycline therapy (without trastuzumab).
* One prior chemotherapy for metastatic breast cancer allowed (may include trastuzumab for HER2+ patients), but no prior Doxil, adriamycin or epirubicin for metastatic breast cancer.
* At least 18 years of age.
* ECOG Performance Status of 0, 1, or 2.
* Adequate organ function including the following:

  * Adequate bone marrow reserve.
  * Cardiac: Left ventricular ejection fraction (LVEF) greater than or equal to 55% by MUGA.
* Negative serum pregnancy test at the time of enrollment for women of child-bearing potential.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments.

Exclusion Criteria:

* Pregnant or nursing women.
* Concurrent anticancer therapy.
* Participation in any investigational drug study within 28 days prior to study entry.
* Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, uncontrolled hypertension, coronary artery disease, congestive heart failure, severe arrhythmia) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
* Symptomatic central nervous system metastases. Patients with asymptomatic brain metastases are allowed. The patient must be stable after radiotherapy for greater than or equal to 2 weeks and off corticosteroids for greater than or equal to 1 week.
* History of interstitial lung disease or pulmonary fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Study Completion 2007-12

PRIMARY OUTCOMES:
Incidence of cardiac toxicity

SECONDARY OUTCOMES:
Objective tumor response rate according to RECIST criteria measured every 2 cycles (every 6 weeks)
Duration of overall response
Time to tumor progression
Progression free survival
Toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Ungerleider, MD, Study Director — Theradex
Locations (25):
- United States (25):
  - New Milford, Connecticut
  - Sharon, Connecticut
  - Torrington, Connecticut
  - Burnsville, Minnesota
  - Edina, Minnesota
  - Maplewood, Minnesota
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Woodbury, Minnesota
  - Columbia, Missouri
  - Albany, New York
  - Amsterdam, New York
  - Hudson, New York
  - Latham, New York
  - Rexford, New York
  - Schenectady, New York
  - Troy, New York
  - Asheville, North Carolina
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Midland, Texas
  - Odessa, Texas
  - Plano, Texas
  - Tyler, Texas